CLINICAL TRIAL: NCT05885633
Title: Phenotypic Components of Polycystic Ovary Syndrome Determine Endometrial Vitamin D Receptor mRNA Expression Pattern
Brief Title: Endometrial Vitamin D Receptor in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Collaborators: Bahçeşehir University (Other); Firat University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UsakUn
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Vitamin D Receptor Defect
Keywords: PCOS; Vitamin D; Endometrium; VD receptor; Hyperandrogenemia; Insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: While the study group consisted of PCOS patients, the control group was selected from non-PCOS patients with male factor infertility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PCOS (Active Comparator): Infertile PCOS patients (n=44)
  Interventions: Procedure: endometrial sampling with pipelle
- Non-PCOS control (Active Comparator): Non-PCOS control with male factor infertility
  Interventions: Procedure: endometrial sampling with pipelle
- Phenotype A (Active Comparator): Phenotype A: HA+OD+PCOM (classical/complete, n=17)
  Interventions: Procedure: endometrial sampling with pipelle
- Phenotype B (Active Comparator): phenotype B: HA+OD (classical/non-PCOM, n=10)
  Interventions: Procedure: endometrial sampling with pipelle
- Phenotype C (Active Comparator): phenotype C: HA+PCOM (ovulatory, n=9)
  Interventions: Procedure: endometrial sampling with pipelle
- Phenotype D (Active Comparator): phenotype D: OD+PCOM (non-hyperandrogenic, n=8).
  Interventions: Procedure: endometrial sampling with pipelle

INTERVENTIONS:
Procedure: endometrial sampling with pipelle — Following oocyte retrieval while the patient was under anesthesia, endometrial tissue sampling was performed with the help of pipelle cannula. A portion of the endometrial tissue was put into RNA stabilization buffer (RNAlater) to be used in qPCR and stored at -20°C until the analysis. The remaining endometrial tissue was first fixed with 10% formalin, followed by paraffin blocking and prepared for immunohistochemical analysis.

SUMMARY:
Vitamin D receptor (VDR) is widely expressed not only in tissues responsible for calcium hemostasis, but also in reproductive organs, including the endometrium. The VDR, which is low in the proliferative phase, starts to increase in the early secretory phase and decreases again in the mid-secretory phase. Enzymes responsible for vitamin d (VD) production and metabolism are expressed locally in the endometrium. Binding of active VD to VDR in nuclear or plasma membrane increases receptivity gene expression and immunomodulators by activating genomic and nongenomic pathways. VDR expression defect has been reported in the decidual cells of recurrent miscarriages. There are no studies investigating the endometrial VDR expression pattern in polycystic ovary syndrome (PCOS) and its phenotypes. The VDR expression pattern in the endometrium of PCOS patients who underwent invitro fertilization /intracytoplasmic sperm injection (IVF/ICSI) and total embryo freezing was analyzed at both mRNA and immunohistochemical. The study group consisted of 44 PCOS patients who were referred to IVF/ICSI because they did not respond to first-line treatment with letrozole or clomiphene citrate (CC). Twenty patients who were scheduled for IVF/ICSI due to male factor infertility and who were matched with the study group in terms of age and body mass index (BMI) were included as the control group. Following egg collection, endometrial tissue was collected by pipelle cannula while the patient was under anesthesia. All good quality blastocysts of both groups were vitrified. The mRNA expression of vitamin D receptor transcript 2 (VDR-X2) and vitamin D receptor transcript 4 (VDR-X4) were determined by quantitative polymerase chain reaction (qPCR). The quantitative cycle equation method was used to calculate the differences between VDR-mRNA expressions. Endometrial VDR and progesterone receptor (PR) immunoreactivity were determined by immunohistochemistry.

DETAILED DESCRIPTION:
Study question: How does the expression of endometrial vitamin D receptor vary according to phenotypes in women with polycystic ovary syndrome (PCOS)?

What is known already: VDR is widely expressed not only in tissues responsible for calcium hemostasis, but also in reproductive organs, including the endometrium. The VDR, which is low in the proliferative phase, starts to increase in the early secretory phase and decreases again in the mid-secretory phase. Enzymes responsible for VD production and metabolism are expressed locally in the endometrium. Binding of active VD to VDR in nuclear or plasma membrane increases receptivity gene expression and immunmodulators by activating genomic and nongenomic pathways. VDR expression defect has been reported in the decidual cells of recurrent miscarriage cases. There are no studies investigating the endometrial VDR expression pattern in PCOS and its phenotypes.

Study design, size, duration: The study group consisted of 44 PCOS patients who were referred to IVF/ICSI because they did not respond to first-line treatment with letrozole or clomiphene citrate (CC). Twenty patients who were scheduled for IVF/ICSI due to male factor infertility and who were matched with the study group in terms of age and BMI were included as the control group. Those who met at least two of the criteria for hyperandrogenemia (HA), ovulatory dysfunction (OD) and polycystic ovarian morphology (PCOM) determined by European Society of Human Reproduction and Embryology/ American Society for Reproductive Medicine were considered PCOS. Following egg collection, endometrial tissue was collected by pipelle cannula while the patient was under anesthesia. All good quality blastocysts of both groups were vitrified.

Participants/materials, setting, methods: The 44 participants in the PCOS group were divided into four phenotypic groups as follows according to the National Institutes of Health (NIH) consensus panel. Phenotype A: HA+OD+PCOM (classical/complete, n=17); phenotype B: HA+OD (classical/non-PCOM, n=10); phenotype C: HA+PCOM (ovulatory, n=9); and phenotype D: OD+PCOM (non-hyperandrogenic, n=8). The mRNA expression of vitamin D receptor transcript 2 (VDR-X2) and vitamin D receptor transcript 4 (VDR-X4) were determined by qPCR. The quantitative cycle equation method was used to calculate the differences between VDR-mRNA expressions. Endometrial VDR and progesterone receptor (PR) immunoreactivity were determined by immunohistochemistry. The histological score formula was used for the quantitative evaluation of VDR and PR immunoreactivity.

Limitations, reasons for caution: The lack of an equal number of participants for each phenotype is our first limitation. Due to the collection of endometrial samples in the IVF/ICSI cycle, the possible effect of ovarian stimulation drugs and the associated increased estrogen levels on the endometrium has not been excluded. Changes in endometrial VDR-mRNA expression could not be confirmed by protein measurement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS
* Approval for IVF/ICSI and total embryo freezing
* Consent to endometrial sampling

Exclusion Criteria:

* Women with hyperandrogenism or ovulatory dysfunction due to non-PCOS etiologies.
* Patients taking vitamin D, insulin sensitizers, lipid-lowering or other hormonal drugs in the last three months were not included.
* Those with a history of mechanical endometrial injury, polypectomy, hysteroscopic myomectomy, endometrioma resection, dilatation/curettage, ovarian drilling and salpingectomy were also excluded.
* Participants with premalignant or malignant endometrial pathology, those with a history of tubal factor infertility, congenital uterine anomaly or any chronic systemic diseases were not included.
* Azoospermia patients were excluded from the study because we preferred ejaculate sperm for ICSI in patients in the control group.

Ages: 26 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — These patients are female patients who are infertile and planned for IVF/ICSI. The condition of being in the reproductive age of the patients was sought.
Enrollment: 64 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
The primary aim of the study was to investigate whether there is a difference in VDR expression in the endometrium of PCOS patients compared to controls by qPCR and immunohistochemical methods | first 3 months
  The VDR expression pattern in the endometrium of PCOS patients who underwent IVF/ICSI and total embryo freezing because they did not respond to first-line ovulation stimulation was analyzed at both mRNA and immunohistochemical levels. Endometrial VDR mRNA expression levels were measured by qPCR method. In addition, samples were stained immunohistochemically to determine the distribution and intensity of VDR in the endometrial tissue. In order to compare the possible relationship between progesterone receptor (PR) distribution and VDR distribution, endometrial samples were also stained immunohistochemically with PR antibody.

SECONDARY OUTCOMES:
To reveal the effects of insulin resistance, HA, OD, and PCOM on endometrial VDR mRNA expression using correlation analyses. | First three months
  Participants in the PCOS group were divided into four groups as phenotype A (HA+OD+PCOM), phenotype B (HA+OD), phenotype C (HA+PCOM) and phenotype D (OD+PCOM) and which phenotypic variable affected VDR mRNA was analyzed.
Clinical pregnancy and miscarriage rates | three months following the first three months
  . Clinical pregnancy was defined as the presence of an intrauterine gestational sac in the transvaginal ultrasonography examination (Clinical pregnancy rate (CPR) = total number of clinical pregnancies/total number of ET cycles × 100%). Fetal loss before 12 weeks of gestation was defined as miscarriage (Miscarriage rate = total number of miscarriages/total number of clinical pregnancies × 100%).

CONTACTS AND LOCATIONS:
Overall Officials: nur DE gungor, assoc. prof., Principal Investigator — BAU IVF-Center; aynur A ersahin, assoc. prof, Principal Investigator — BAU IVF-Center; arzu yurci, assoc. prof., Principal Investigator — Memorial IVF-Center; Ulun ulug, prof, Principal Investigator — Halic University; meltem yardım, specialist, Principal Investigator — Yerkoy State Hospital; nilufer celik, assoc. prof., Principal Investigator — Dr. Behcet Uz Children's Hospital; ahmet tektemur, assoc. prof, Principal Investigator — Firat University; Tuncay Kuloglu, Assoc. prof, Principal Investigator — Firat University; Kagan Gungor, Assoc. prof, Principal Investigator — Medeniyet University
Locations (1):
- Usak University Training and Research Hospital, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Carmina E, Longo RA. Increased Prevalence of Elevated DHEAS in PCOS Women with Non-Classic (B or C) Phenotypes: A Retrospective Analysis in Patients Aged 20 to 29 Years. Cells. 2022 Oct 17;11(20):3255. doi: 10.3390/cells11203255. PMID 36291122